CLINICAL TRIAL: NCT04842799
Title: BRCA-DIRECT: Randomised Evaluation in Women Diagnosed With Breast Cancer of Digitally-delivered Pre-test Information for BRCA-testing
Brief Title: Digital Delivery of Information About Genetic Testing for Breast Cancer
Acronym: BRCA-DIRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: University of Sussex (Other); University of Manchester (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CCR5234; C61296/A29423 (Other Grant/Funding Number: Cancer Research UK); 47406 (Registry Identifier: CPMS ID)
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Neoplasm Female
Keywords: Genetic Testing; Digital Intervention

STUDY DESIGN:
Intervention Model Description: Participants are initially randomised 1:1 to receive genetic pre-test information either via the BRCA-DIRECT digital platform or a genetic counselling telephone appointment. Once the participants BRCA-gene test result becomes available, they are then randomised sequentially depending on the result of the genetic test. Participants with a negative (normal) result are randomised to receive this information either via the BRCA-DIRECT digital platform or a genetic counselling telephone appointment. Participants with a positive result will not be randomised and instead will always have a genetic counselling telephone appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Digital delivery of genetic pre-test information (Experimental): Half of participants will be provided with genetic pre-test information via the BRCA-DIRECT digital platform.
  Interventions: Other: Digital Delivery of Pre-Genetic Testing Information via the BRCA-DIRECT Platform
- Genetic counselling telephone appointment to discuss genetic pre-test information (No Intervention): Half of participants will be provided with genetic pre-test information via the normal standard pathway - a telephone consultation with a Genetic Counsellor.
- Digital delivery of BRCA-gene testing results (Experimental): 97.5% of participant's with a negative (normal) result will receive their BRCA-gene testing result via the BRCA-DIRECT digital platform.
  Interventions: Other: Digital Delivery of Genetic Test Results via the BRCA-DIRECT Platform
- Genetic counselling telephone appointment to discuss BRCA-gene testing results (No Intervention): 2.5% of participants with a negative (normal) result and those with positive results will receive their BRCA-gene testing result via the normal standard pathway - a telephone consultation with a Genetic Counsellor.

INTERVENTIONS:
Other: Digital Delivery of Pre-Genetic Testing Information via the BRCA-DIRECT Platform — Participants will receive a link to the digital pre-test information. This will consist of text covering: Genetics and cancer risk; Genetics testing; What will happen if your test is positive; What will happen if your test is negative; Implications for insurance.
  Where relevant, parts of the text will be linked through to additional information, such as insurance advice from the Association of British Insurers. Participants will be able to call a genetic counsellor on the hotline during weekday office hours, should they have any questions or require further information.
  Arms: Digital delivery of genetic pre-test information
Other: Digital Delivery of Genetic Test Results via the BRCA-DIRECT Platform — Participants will receive a digital message that their results are available. When they click this, they will receive digital notification of their negative (normal) result in short form. Full details will be provided in an individualised letter.
  Arms: Digital delivery of BRCA-gene testing results

SUMMARY:
BRCA-DIRECT is a pragmatic, randomised, non-inferiority evaluation that aims to evaluate whether digital delivery of pre-test information for BRCA-testing in breast cancer patients is non-inferior to current standard practice of 1:1 delivery from a healthcare professional as measured by rate of uptake of the genetic testing.

DETAILED DESCRIPTION:
Participants will be recruited via breast clinics in two oncology centres. Patients will be provided with a study pack containing information about the study. If in clinic, the patient can complete an expression of interest form and a saliva/blood sample will be stored until consent to the study is received. The consent form and saliva sample can be completed at home and sent to the study team.

On receipt of a signed study consent form, the local site will confirm the patient's eligibility and enter details required for study conduct onto the BRCA-DIRECT databases.

After 24 hours, the participant will be sent a link to the BRCA-DIRECT study platform interface. This link enables the participant to progress through the study or withdraw if they have changed their mind.

Participants will be randomised 1:1 to receive either:

1. Telephone consultation with a genetic counsellor (standard of care) The telephone consultations will be as per standard practice of the qualified genetic counsellor delivering the pre-test information.
2. Digital delivery of pre-test information via BRCA-DIRECT platform (intervention)

Participants will receive a link to the digital pre-test information. This will consist of text covering:

* Genetics and cancer risk
* Genetics testing
* What will happen if your test is positive
* What will happen if your test is negative
* Implications for insurance

All participants will have access to a Genetic Counsellor hotline at all stages of the process.

For both arms, if a participant decides to proceed with the genetic test they will sign a digital 'BRCA-test consent' form, which will be formatted to BSGM (British Society of Genomic Medicine) standards. All participants will receive a copy of their signed BRCA-test consent form via secure email/post. The participant will have two days following test-consent to reverse the decision to proceed with the BRCA-test. Beyond those two days, the test will proceed.

The laboratory testing is a standard UK NHS (National Health Service) genetic test. This is delivered for both the intervention arm and the standard-of-care arm.

Participants with a negative (normal) genetic test result will be randomised to receive results either digitally, or via telephone consultation with the Genetic Counsellor. Any individuals with a positive result will receive their result by telephone. Following delivery of results, a results letter and copy of the pathology report will be sent to the participant and their medical team.

The participants will be invited to complete Quality of Life questionnaires, a knowledge test and satisfaction survey at various time points throughout the study via the BRCA-DIRECT platform.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive breast cancer or high-grade ductal carcinoma in situ (DCIS)
* Female
* Aged 18 years or over
* Access to smartphone or email + internet
* Good comprehension of the English Language

Exclusion Criteria:

• Previous testing for BRCA1/2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Uptake of genetic testing | From the point the participant completes the initial Expression of Interest form at Enrolment, until the participant completes the BRCA-test consent approx. 1-3 weeks later.
  Proportion of patients proceeding with the BRCA-gene test following receipt of pre-test information

SECONDARY OUTCOMES:
Knowledge about genetic testing for BRCA genes | 7 days after the BRCA-test consent has been signed the patient will complete the Knowledge Questionnaire
  Test participant knowledge following delivery of pre-test information via a Knowledge Questionnaire (study specific) of 12 True/False/Unsure questions for a total possible score of 12/12.
Anxiety following delivery of pre-test information and test results by the Spielberger State-Trait anxiety inventory | The participant completes Quality of Life Questionnaires at baseline, 7 days after BRCA-test consent and then at 7 and 28 days after the notification that the patients BRCA-test results are available
  Participant Quality of Life Questionnaire scores collected before pre-test information and after test results received. The Spielberger state-trait anxiety inventory (STAI) consists of two self-administered, 20-item questionnaires, with each item rated on a four-point Likert scale. It assesses anxiety proneness (trait) and the current state of anxiety change (state). The Trait anxiety is measured only once before pre-test information, and the State at each time point. High STAI scores signify greater anxiety.
Assessment of number of participants who uptake of digital genetic testing | The point at enrolment where the participant completes the initial expression of interest form
  Potential participant decline on account of lack of digital access
'Test-offer-to-results' time | The point at enrolment where the participant completes the expression of interest form until the notification that the patients BRCA-test results are available (approx. 6-8 weeks)
  To compare 'Test-offer-to-results' time of the BRCA-DIRECT digital model compared to an audit of timings under current pathways at participating centres
Helpline usage | The point at which a participant who has been randomised to digital delivery of pre-test information contacts the telephone helpline, between date of randomisation and date of participant withdrawal/study completion 28 days after receiving test results
  Evaluate proportion of patients receiving digital pre-test information who require 1:1 discussion via the helpline
Healthcare professional satisfaction | Healthcare professional completes the Healthcare Professional Feedback Survey after interacting with the study, following completion of all patients through the study (approximately 14 months from study recruitment start).
  Healthcare Professional Feedback Survey completion to evaluate how satisfied Healthcare professionals were with the BRCA-DIRECT digital model
Patient satisfaction | 7 days after the notification that the patients BRCA-test results are available the participant completes the Participant Satisfaction Survey
  Participant Satisfaction Survey (study specific) completion to evaluate how satisfied patients were with the BRCA-DIRECT digital model, consisting of 9 questions, of which 3 are ranked on a scale of 1-5 (1 - not satisfied to 5 - very satisfied) and others are multi-choice.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Evans, Principal Investigator — Manchester University NHS Foundation Trust; Angela George, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Wythenshawe Hospital, Manchester, England
  - Royal Marsden Hospital, Chelsea, Chelsea, London
  - Royal Marsden Hospital, Kingston, Kingston, London
  - Royal Marsden Hospital, Sutton, Sutton, Surrey
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torr B, Jones C, Choi S, Allen S, Kavanaugh G, Hamill M, Garrett A, MacMahon S, Loong L, Reay A, Yuan L, Valganon Petrizan M, Monson K, Perry N, Fallowfield L, Jenkins V, Gold R, Taylor A, Gabe R, Wiggins J, Lucassen A, Manchanda R, Gandhi A, George A, Hubank M, Kemp Z, Evans DG, Bremner S, Turnbull C. A digital pathway for genetic testing in UK NHS patients with cancer: BRCA-DIRECT randomised study internal pilot. J Med Genet. 2022 Dec;59(12):1179-1188. doi: 10.1136/jmg-2022-108655. Epub 2022 Jul 22. PMID 35868849
- [Derived] Torr B, Jones C, Kavanaugh G, Hamill M, Allen S, Choi S, Garrett A, Valganon-Petrizan M, MacMahon S, Yuan L, Way R, Harder H, Gold R, Taylor A, Gabe R, Lucassen A, Manchanda R, Fallowfield L, Jenkins V, Gandhi A, Evans DG, George A, Hubank M, Kemp Z, Bremner S, Turnbull C. BRCA-DIRECT digital pathway for diagnostic germline genetic testing within a UK breast oncology setting: a randomised, non-inferiority trial. Br J Cancer. 2024 Nov;131(9):1506-1515. doi: 10.1038/s41416-024-02832-2. Epub 2024 Oct 1. PMID 39349619
- See also: A digital pathway for genetic testing in UK NHS patients with cancer: BRCA-DIRECT randomised study internal pilot (publication of pilot phase study data for the first 130 participants recruited) — https://pubmed.ncbi.nlm.nih.gov/35868849/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04842799/Prot_SAP_000.pdf